CLINICAL TRIAL: NCT02518763
Title: Vitamin D Supplementation in Postmenopausal Women With Osteoporosis: Proposal of a Therapeutic Regimen in Practice
Acronym: VITAD
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-090
Record Dates: First submitted 2015-08-06; First posted 2015-08-10 (Estimated); Last update posted 2015-08-10 (Estimated); Status verified 2015-08

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis | interventions — Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vitamin D3, 100 000 IU weekly, 4 times (Experimental)
  Interventions: Drug: Vitamin D3, 100 000 IU weekly, 4 times; Biological: 25 OH vitamin D serum concentration measurements

INTERVENTIONS:
Drug: Vitamin D3, 100 000 IU weekly, 4 times
Biological: 25 OH vitamin D serum concentration measurements

SUMMARY:
The vitamin D deficiency (25OHD) is very common and affects about 80% of the population of French osteoporotic women over 50 years [5]. It contributes significantly to bone fragility and consequently the risk of fracture. To remedy this deficit, it is necessary to provide a suitable and sustainable supplementation. Changes in vitamin D deficiency ranging from undetectable to a 25OHD value very close to 30ng / ml lead to differences in therapeutic regimens, specific to each clinician in the absence of precise data in the literature. No consensus on supplementation dosages and methods have been proposed so far. Also, given the frequency of vitamin D deficiency including osteoporosis observed in the population, it became necessary to establish a single, uniform regimen for all patients with osteoporosis

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women ≥ 50 years
* Osteoporosis with BMD T-score ≤ -2.7DS -2.5DS to at least one of the two main sites analyzed, with or without fracture
* having signed an informed consent

Exclusion Criteria:

* Taking a "loading dose" of vitamin D in the last six months (a daily intake in combination with calcium will not be a cause of exclusion but should be discontinued during the study).
* Taking an osteoporosis treatment combined with vitamin D in the same tablet (or Adrovance Fosavance * *)
* Treatment with thiazide diuretic
* Known malabsorption (celiac disease)
* Scalable Endocrine disorders: hyperthyroidism, hyperparathyroidism, hypoparathyroidism.
* Persistent or nephrolithiasis occurred in the previous 5 years
* known sarcoidosis
* Persons under guardianship or trusteeship
* Hypercalcemia and hypercalciuria
* 25OH vitamin D levels> 50ng / ml

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2011-06; Primary Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Serum 25 OH vitamin D concentration | 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Caen, France